CLINICAL TRIAL: NCT03454139
Title: A Comparison of Perioperative Analgesic Effects of Preemptive Subcostal Transversus Abdominis Plane (TAP) Block and Paracetamol for Percutaneous Nephrolithotomy
Brief Title: Subcostal TAP Block For Percutaneous Nephrolithotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Guniz M.Koksal, Clinical Professor, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 186
Record Dates: First submitted 2018-02-12; First posted 2018-03-05 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Nephrolithiasis
Keywords: percutaneous nephrolithotomy; subcostal transversus abdominis plane block; pain; paracetamol; tramadol; morphine; nephrolithiasis; lidocaine; bupivacaine
MeSH Terms: conditions — Nephrolithiasis; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (2):
- Subcostal TAP group (Active Comparator): Ultrasound guided Subcostal transversus abdominis plane block is performed after anesthesia induction and endotracheal intubation , to the side where kidney stone is. A composition of 10 ml Lidocaine %1 plus 10 ml physiologic saline solution plus 10 ml Bupivacaine %0,25 , total of 30 ml of local anesthetic mixture is administered into the area between internal oblique muscle fascia and transversus abdominis muscle fascia. After that, the patient is positioned to lithotomy position and the open-end catheter is inserted. After that the patient is turned to prone position and the percutaneous nephrolithotomy is performed. Tramadol 100 mg iv is administrated 20 minutes before the end of the surgery. Morphine patient controlled analgesia is planned for postoperative pain management.
  Interventions: Procedure: Subcostal transversus abdominis plane block
- Non- TAP group (No Intervention): Percutaneous nephrolithotomy is performed under general anesthesia. No regional analgesia is administered to this patients. Paracetamol 1000 mg/100ml; iv and Tramadol 100mg iv is administered 20 minutes before the end of the surgery for postoperative analgesia. Morphine patient controlled analgesia is planned for postoperative pain management.

INTERVENTIONS:
Procedure: Subcostal transversus abdominis plane block — Ultrasound guided Subcostal transversus abdominis plane block is performed after anesthesia induction and endotracheal intubation , to the side where kidney stone is. A composition of 10 ml Lidocaine %1 plus 10 ml physiologic saline solution plus 10 ml Bupivacaine %0,5 , total of 30 ml of local anesthetic mixture is administered into the area between internal oblique muscle fascia and transversus abdominis muscle fascia.
  Arms: Subcostal TAP group

SUMMARY:
Percutaneous nephrolithotomy (PCNL) is a minimally- invasive procedure for removing kidney stones. The small incision of PCNL is performed medially from the posterior axillary line according to stones location. Despite the small skin incision patients suffer from postoperative pain due to visceral pain and intercostal nerve injury. The aim of this study is to evaluate the perioperative analgesic effect of subcostal transversus abdominis plane (TAP) block performed prior to PCNL procedure.

Primary outcome of our study was Morphine consumption at 48th hour after the surgery. Secondary outcomes were perioperative fentanyl consumption; postoperative Verbal Analog Scale and additional analgesic drug requirement.

DETAILED DESCRIPTION:
Patients who were scheduled for elective percutaneous nephrolithotomy were randomized into two groups: Group TAP and Group IV. General anesthesia was induced with propofol 2 mg/kg, fentanyl 1 mcgr/kg and rocuronium 0,6 mg/kg and maintained with sevoflurane 2% in 40%:60% oxygen/air mixture and fentanyl 0,5 mcgr/kg and rocuronium 10 mg, if necessary. Unilateral Transversus abdominis plane block was performed with total of 30 ml volume of local anesthetic solution (20ml Bupivacaine 0,125% and 10ml Lidocaine 1%) after intubation but before surgery to the Group TAP patients. Paracetamol 1 gr, iv was given to the Group IV 20 minutes before the end of the surgery. Also 100mg Tramadol,iv was administered 20 minutes before the end of the surgery to the both groups. Morphine iv patient controlled analgesia was applied to both groups. Perioperative fentanyl consumption; postoperative Verbal Analog Scale, morphine consumption and additional analgesic drug requirement were determined. Data of perioperative complications and adverse effects were also collected. Chi square with Yates correction and Mann Whitney U tests were used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* patients enrolled for percutaneous nephrolithotomy (PCNL) surgery
* ASA (American Society of Anesthesiologists) score I-III

Exclusion Criteria:

* patients with chronic pain
* patients on opioid or other analgesic drugs
* BMI (body mass index) higher than 40
* allergies for drugs used in the study
* chronic renal failure receiving dialysis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-10; Primary Completion 2017-07 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Total morphine used (milligram) | 48 hours after the end of the surgery
  Morphine patient controlled analgesia (PCA) is applied for both patient groups. PCA settings are bolus: 1 mg Morphine and lock time:10 minutes.

SECONDARY OUTCOMES:
Morphine consumption (milligram) | 1- 0 minutes; 2- 30 minutes; 3- 1 hour; 4- 2 hours; 5- 3 hours; 6- 12 hours; 7- 24 hours; 8- 48 hours after the end of the surgery
  Morphine patient controlled analgesia (PCA) is applied for both patient groups. PCA settings are bolus: 1 mg Morphine and lock time:10 minutes.
Additional analgesic requirement | 1- 0 minutes; 2- 30 minutes; 3- 1 hour; 4- 2 hours; 5- 3 hours; 6- 12 hours; 7- 24 hours; 8- 48 hours after the end of the surgery
  Additional analgesia regimen is planned as (in order of administration): 1000 mg/100ml Paracetamol iv infusion; 50 mg Dexketoprofen trometamol iv; 100mg Tramadol iv infusion. Additional analgesia is administrated when VAS is equal to or higher than 4.
Visual Analog Scale (VAS) | 1- 0 minutes; 2- 30 minutes; 3- 1 hour; 4- 2 hours; 5- 3 hours; 6- 12 hours; 7- 24 hours; 8- 48 hours after the end of the surgery
  Patients are asked to rate their pain according to 10 point VAS in which 0 means "no pain at all" , 10 means "worst pain ever".
Fentanyl consumption (microgram/kg) | 0 minute after the end of the surgery
  Fentanyl 1 microgram/kg is administered at anesthesia induction. Fentanyl 0,5 microgram/kg is added during the surgery, if needed (20% increasing of heart rate or mean blood pressure)